CLINICAL TRIAL: NCT04643886
Title: A Multicenter, Open-label, Multiple Dose Study in Patients With Geographic Atrophy Secondary to Dry Age-related Macular Degeneration to Evaluate the Safety, Tolerability, Pharmacodynamics, and Immunogenicity of Repeat Intravitreal Injections of GEM103
Brief Title: A Multiple Dose Study of Repeat Intravitreal Injections of GEM103 in Dry Age-related Macular Degeneration
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: no further benefit
Sponsor: Gemini Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEM-CL-10302; REGATTA (Other: Gemini Therapeutics)
Record Dates: First submitted 2020-11-16; First posted 2020-11-25 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Dry Age-related Macular Degeneration; Geographic Atrophy; Macular Degeneration; Retinal Disease; Retinal Degeneration
MeSH Terms: conditions — Geographic Atrophy; Macular Degeneration; Retinal Diseases; Retinal Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort with Genetic Profile A (Experimental): Subjects will have Genetic Profile A.
  Intervention: Biological: GEM103.
  Interventions: Drug: GEM103
- Cohort with Genetic Profile B (Experimental): Subjects will have Genetic Profile B.
  Intervention: Biological: GEM103
  Interventions: Drug: GEM103

INTERVENTIONS:
Drug: GEM103 — Biological

SUMMARY:
This study is designed to investigate the safety, PK/PD, biomarker and early clinical effects of repeat GEM103 IVT injections.

DETAILED DESCRIPTION:
This is a Phase 2a, multi-center, open-label, multiple dose study in subjects with geographic atrophy (GA) secondary to dry Age-related Macular Degeneration (dry AMD) to investigate the safety, PK/PD, biomarker and early clinical effect of GEM103 repeat IVT injections.

Subjects will undergo clinical and ophthalmic assessments for determination of inclusion in the study. Subjects who participated in the Phase 1 Study (GEM-CL-10301) as well as treatment naïve subjects that did not participate in the GEM-CL-10301 Study and who meet all eligibility criteria will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. At least 50 years old at the time of signed informed consent.
2. Must have one of the following genetic profiles:

   1. Genetic Profile A.
   2. Genetic Profile B.
3. BCVA in the study eye of 24 to 83 letters using ETDRS Chart Visual Acuity (VA) Scale (approximately equivalent to Snellen VA of 20/25 to 20/320).
4. Confirmed diagnosis of GA in the study eye where total size of all GA lesions in the study eye must be within 0.5 to 15.01- and 7- disc areas.
5. Sufficiently clear ocular media and able to cooperate with ophthalmic visual function testing and anatomic assessment in the study eye.
6. Understands the full nature and purpose of the study and provides informed consent prior to initiation of any study procedure; all subjects with a reproductive potential must agree to use effective contraceptive methods through the end of study (EOS) Visit.

Exclusion Criteria:

1. Presence of the following ocular conditions - in the study eye:

   1. Any history of exudative Age-related Macular Degeneration or choroidal neovascularization.
   2. Any active ocular disease or condition that could confound the assessment of the macula or be a contraindication to IVT injection.
   3. Any intraocular surgery, with the exception of stable intraocular lens replacement surgery more than 3 months prior to consent.
   4. Aphakia or complete absence of the posterior capsule.
   5. History of laser therapy to the macula or fundus or extensive laser to the retina.
   6. Prior corneal transplant.
2. Presence of any of the following ocular conditions - in either eye:

   1. History of herpetic infection.
   2. Concurrent disease that could require medical or surgical intervention during the study period.
   3. Active uveitis and/or vitritis (grade: trace or above).
   4. History of idiopathic or autoimmune-associated uveitis.
   5. Active blepharitis, conjunctivitis, keratitis, episcleritis, scleritis, or endophthalmitis.
   6. Any ophthalmologic condition that reduces the clarity of the media and that, in the opinion of the Investigator, interferes with ophthalmologic examination.
3. In the opinion of the Investigator, the subject has any prior or ongoing medical condition (e.g., ocular other than dry AMD, systemic, psychiatric) or clinically significant screening laboratory value that may present a safety risk, interfere with study compliance or study follow-up, or confound data interpretation throughout the follow-up period.
4. Female subjects must not be pregnant or lactating, nor plan to become pregnant during the study.
5. Current use of medications known to be toxic to the lens, retina, or optic nerve.
6. Use of any investigational new drug or other experimental treatment in the last 6 months, and/or receipt of any prior gene therapy (e.g., AAV) or ocular device implantation (other than PCIOL placement following cataract surgery)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Safety of intravitreal (IVT) injections of GEM103, as measured by number of subjects with ocular adverse events. | 18 months

SECONDARY OUTCOMES:
To describe the clinical effect of GEM103 IVT injection, as the change from baseline in best corrected visual acuity (BCVA) scores as assessed by ETDRS scale. | 6 months
To evaluate the total CFH levels in aqueous humor after GEM103 IVT injection, whenever possible. | 6 months

CONTACTS AND LOCATIONS:
Locations (29):
- United States (29):
  - Gemini Clinical Trial Site, Phoenix, Arizona
  - Gemini Clinical Trial Site, Bakersfield, California
  - Gemini Clinical Trial Site, Beverly Hills, California
  - Gemini Clinical Trial Site, Oxnard, California
  - Gemini Clinical Trial Site, Poway, California
  - Gemini Clinical Trial Site, Santa Barbara, California
  - Gemini Clinical Trial Site, Santa Maria, California
  - Gemini Clinical Trial Site, Golden, Colorado
  - Gemini Clinical Trial Site, New London, Connecticut
  - Gemini Clinical Trial Site, Palm Beach Gardens, Florida
  - Gemini Clinical Trial Site, St. Petersburg, Florida
  - Gemini Clinical Trial Site, Tallahassee, Florida
  - Gemini Clinical Trial Site, Winter Haven, Florida
  - Gemini Clinical Trial Site, Augusta, Georgia
  - Gemini Clinical Trial Site, Marietta, Georgia
  - Gemini Clinical Trial Site, Oak Park, Illinois
  - Gemini Clinical Trial Site, Indianapolis, Indiana
  - Gemini Clinical Trial Site, Chesterfield, Missouri
  - Gemini Clinical Trial Site, St Louis, Missouri
  - Gemini Clinical Trial Site, Reno, Nevada
  - Gemini Clinical Trial Site, Bloomfield, New Jersey
  - Gemini Clinical Trial Site, Asheville, North Carolina
  - Gemini Clinical Trial Site, Charlotte, North Carolina
  - Gemini Clinical Trial Site, Eugene, Oregon
  - Gemini Clinical Trial Site, Rapid City, South Dakota
  - Gemini Clinical Trial Site, Abilene, Texas
  - Gemini Clinical Trial Site, Dallas, Texas
  - Gemini Clinical Trial Site, The Woodlands, Texas
  - Gemini Clinical Trial Site, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tzoumas N, Riding G, Williams MA, Steel DH. Complement inhibitors for age-related macular degeneration. Cochrane Database Syst Rev. 2023 Jun 14;6(6):CD009300. doi: 10.1002/14651858.CD009300.pub3. PMID 37314061